CLINICAL TRIAL: NCT03884959
Title: A Prospective, Open Label, Safety and Efficacy Study of Infusions of HepaStem in Urea Cycle Disorders Pediatric Patients
Brief Title: A Safety and Efficacy Study of Infusions of HepaStem in Urea Cycle Disorders Pediatric Patients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decided to stop enrollment
Sponsor: HLB Cell Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HEP002KR
Record Dates: First submitted 2019-03-03; First posted 2019-03-21 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-02

CONDITIONS: Urea Cycle Disorder
Keywords: Urea Cycle Disorder; Hyperammonemia; Metabolic Decompensation
MeSH Terms: conditions — Urea Cycle Disorders, Inborn; Hyperammonemia

STUDY DESIGN:
Intervention Model Description: This is a single group, open label study
Masking Description: No Masking applied.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HepaStem Infusion (Experimental): A calculated dose based on patient's body weight will be administered via Permanent mesenteric Portal Access and Catheter for four times or a Transient Percutaneous Transhepatic Catheter for three times.
  Interventions: Biological: HepaStem Infusion

INTERVENTIONS:
Biological: HepaStem Infusion — HepaStem will be infused intravenously into the portal vein, either (1) via a permanent mesenteric PAC inserted surgically in an affluent of the portal vein; or (2) through a transient percutaneous transhepatic catheter inserted in to the portal vein under radio guidance.

SUMMARY:
This is a phase2, prospective, open label study designed to investigate the safety and efficacy of several infusions of HepaStem. This study will include 5 pediatric Urea Cycle Disorder (UCD) patients under 12 years old.

Its assessment includes all safety parameters and an efficacy assessment based on 13C tracer tests, ammonia, medication and diet changes.

HepaStem will be administered in addition to the conventional UCD treatments.

DETAILED DESCRIPTION:
Patient eligibility will be assessed during the Screening visit. The investigator should ensure that the chronic metabolic treatment (i.e. balance between low protein diet, supplements in amino acid mix, nitrogen scavenger and supplements in arginine and/or citrulline) of the patient is optimized for his/her metabolic condition.

During the baseline period, 3 study visits will take place at 6 weeks interval for assessing the metabolic condition and the chronic metabolic treatment of the patient.

A calculated dose based on patient's body weight will be administered via Permanent mesenteric Portal Access and Catheter for four times or a Transient Percutaneous Transhepatic Catheter for three times.

The follow-up period will start approximately 12 weeks after the first HepaStem infusion day. This period will last approximately 9 months. Study visits will take place every 1.5month, FU visit 1 to FU visit 7.

Primary Objective:

1. To demonstrate the functional efficacy of HepaStem at 6 months after initiation of infusion in terms of ureagenesis improvement based on a functional test (13C tracer method)
2. To evaluate the safety of Hepastem up to one year after initiation the Hepastem infusion

Secondary Objective:

1. To evaluate the efficacy of Hepastem in terms of functional, clinical, and biochemical parameters up to one year after initiation of the infusion.

ELIGIBILITY:
Inclusion Criteria:

* The patient is a pediatric patient <12 years
* The patients presents with one of the following UCDs. (CPS1D, OTCD, ASSD, ASLD, ARGD)
* The patient has severe disease with impaired protein tolerance defined as: chronic protein restricted diet AND chronic treatment with at lease one nitrogen scavenger.
* The patient shows patency of the portal vein and its branches including mesenteric veins, with normal flow velocity as confirmed by Doppler US and accessibility of the portal vein and/or affluents.
* The patient (if capable of signing) and parents or legal representative have signed a written informed consent form.

Exclusion Criteria:

* The patient presents acute liver failure.
* The patient presents clinical or radiological evidence of liver cirrhosis.
* The patient presents or has a history of hepatic or extrahepatic malignancy.
* The patient has a known clinically significant cardiac malformation.
* The patient has a personal history of venous thrombosis, or has a clinically significant abnormal value for protein S, protein C, anti-thrombin III, and/or activated Protein C Resistance (aPCR) at screening. In case of known family history, a complete coagulation work-up should be performed. in all above described cases, results need to be discussed with sponsor before enrolling the patient in the study.
* Patient currently receiving other unapproved investigational drug or device.
* The patient underwent previous mature liver cell or stem cell transplantation or received an organ liver transplant or received HepaStem infusion.
* The patient has a contraindication to methylprednisolone, tacrolimus.
* The patient has a known hypersensitivity or allergy to heparin.
* The patient has a known hypersensitivity or allergy to the antibiotics preventing post-operative infections that are prescribed according to institutional guidelines, and no alternative prophylaxis can be found.
* The patient had or has a renal insufficiency treated by dialysis.
* The patient requires valproate therapy.
* The patient has a known hypersensitivity or allergy to contrast agents (if applicable) that cannot be treated adequately.
* The patient has a thrombosis of the portal vein or persisting impairment of anterograde portal blood flow.
* The patient has a porto systemic shunt or fistula assessed by Doppler US or an Arantius channel or protal hypertension.
* The site where the catheter is intended to be placed has previously suffered from venous thrombosis or vascular surgical procedures.
* The patient has an ongoing infection or suffered from an infection in the last 2 weeks (including active EBV infection at screening). The patient may be enrolled after resolution of the infection.
* There is any significant condition or disability that, in the investigator's opinion, may interfere with the patient's participation in the study.

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2020-11-04 (Actual); Study Completion 2020-11-04 (Actual)

PRIMARY OUTCOMES:
Change of ureagenesis | at 6 months after the first infusion
  Change of de novo ureagenesis at 6 months after the first infusion:
  absolute 13C blood urea AUC-120 min quantified with the 13C Tracer method at FU visit 3 compared with baseline evaluations.
Hemodynamics (measurement of portal vein pressures) | up to 12 months after the first infusion
  Safety evaluation in terms of portal-vein hemodynamics
Number of subjects with anti-HLA antibody | up to 12 months after the first infusion
  Safety evaluation in terms of de novo detection of donor-specific circulating anti-HLA antibodies and/or other immune-related markers
Number of subjects with SAEs and AEs | up to 12 months after the first infusion
  Safety evaluations in terms of SAEs and clinically significant AEs related to study procedures

SECONDARY OUTCOMES:
Change of ureagenesis | at 3, 9 and 12 months after the first infusion
  Change of de novo ureagenesis at 3, 9 and 12 months after the first infusion:
  absolute 13C blood urea AUC-120 min quantified with the 13C Tracer method at FU visit 1, 5 and 7 compared with baseline evaluations.
Change of chronic protein intake | Up to 12 months after the first infusion
  Chronic protein intake (total and natural protein, reported in mg/kg/day and reported as compared to WHO safe level for age) considering diet evaluations at study visits during baseline period and at scheduled study visits during the follow-up period.
Change of chronic nitrogen scavenger dose | Up to 12 months after the first infusion
  Chronic nitrogen scavenger dose (mg/kg/day) considering reported doses at scheduled study visits during baseline period and at scheduled study visits during the follow-up period.
Change of the level of blood ammonia | Up to 12 months after the first infusion
  Blood ammonia considering values measured at scheduled study visits during screening and baseline periods ant at scheduled study visits during the follow-up period.
Change of relevant blood amino acids values | Up to 12 months after the first infusion
  Relevant blood amino acids considering values measured at scheduled study visits during the screening and baseline periods and at scheduled study visits during the follow-up period.
Number of subjects with Metabolic decompensations | Up to 12 months after the first infusion
  Metabolic decompensations (hyperammonemia episodes with evocative symptomatology such as drowsiness, gastrointestinal symptoms and treated at hospital), considering all collected events during screening and baseline periods, during active treatment period, during follow-up period.
Change of chronic single amino acid intake | Up to 12 months after the first infusion
  Chronic single animo acid intake considering reported doses at study visits during baseline period and at study visits during the follow-up period.
Evaluation of cognitive skill | Up to 12 months after the first infusion
  Change of patient's cognitive skill score between the baseline period (at Baseline visit 1) and the follow-up period (at Follow up visit 7) will be evaluated by the Bayley Scales of Infant Development. (7 classes, from extremely low to very superior)
Evaluation of Behavior indicator | Up to 12 months after the first infusion
  Behavior indicator will be evaluated by the Child Behavior Checklist (CBCL) at Baseline visit 1, during follow-up period at 4.5 months, 7.5 months and 12 months post-first fusion (at Follow up visit 2, 4, 7)
Evaluation of health-related Quality of Life (QoL) indicator | Up to 12 months after the first infusion
  Health-related QoL indicator will be evaluated by the Pediatric Quality of Life Inventory at Baseline visit 1, during follow-up period at 4.5 months, 7.5 months and 12 months post-first fusion (at Follow up visit 2, 4, 7)

CONTACTS AND LOCATIONS:
Overall Officials: Sanghoon Lee, MD. Ph.D, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea